CLINICAL TRIAL: NCT02687360
Title: Imaging the Effects of rTMS on Chronic Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: funding not received
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Diana Martinez, Professor of Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7208
Record Dates: First submitted 2015-12-23; First posted 2016-02-22 (Estimated); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain; Opioid-use Disorder
Keywords: Methadone
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active rTMS stimulation (Active Comparator): This arm will receive high-frequency rTMS pulses directed at the medial prefrontal and anterior cingulate cortices.
  Interventions: Device: Active rTMS treatment
- Sham rTMS stimulation (Sham Comparator): The sham coil setting is designed to mimic the auditory artifact and the scalp sensations evoked by the real coil and to produce activation of facial muscles similar to the effect of active rTMS without stimulating the brain itself.
  Interventions: Device: Sham rTMS treatment

INTERVENTIONS:
Device: Active rTMS treatment — In the active treatment, magnetic power output will be delivered to the participants through the coils.
  Other Names: rTMS
  Arms: Active rTMS stimulation
Device: Sham rTMS treatment — The sham coil setting is designed to mimic the auditory artifact and the scalp sensations evoked by the real coil, and to produce activation of facial muscles similar to the effect of a real H coil, without stimulating the brain itself.
  Arms: Sham rTMS stimulation

SUMMARY:
Chronic pain is highly prevalent in patients with opioid use disorder on methadone maintenance therapy, and associated with problems related to psychosocial functioning, medical and psychiatric health, and substance craving and use. Neuroimaging has strongly correlated pain processing with the medial prefrontal and dorsal anterior cingulate cortices. This study will investigate the effects of repetitive transcranial magnetic stimulation (rTMS) using the H7 coil targeting these same brain areas for the treatment of chronic pain in patients on methadone maintenance therapy,and magnetic resonance imaging and spectroscopy (MRI/MRS) will be used to evaluate target engagement and mechanism.

DETAILED DESCRIPTION:
The research aims of this study are to (1) investigate the efficacy of repetitive transcranial magnetic stimulation (rTMS) of the medial prefrontal cortex and dorsal anterior cingulate cortex for the treatment of chronic non-cancer pain in participants with opioid use disorder on methadone-maintenance therapy, and (2) investigate target engagement by measuring changes in gray matter volume and glutamate-glutamine in these brain regions by magnetic resonance imaging and spectroscopy. Given the high incidence of chronic pain in the OUD population and specifically the methadone-maintained population, there is great need for effective treatments. Untreated chronic pain contributes to medical and psychiatric problems, reduced quality of life, and increased risk of substance use and overdose. Non-invasive neuromodulation like rTMS, which is currently FDA-approved for treatment-resistant depression and OCD, holds promise as a safe and effective therapeutic. This project will investigate rTMS of brain regions known to process the affective and cognitive components of chronic pain, utilizing a treatment protocol modeled after the FDA-approved protocol for obsessive-compulsive disorder.

Volunteers will be randomized in a double-blind manner to 25 sessions (5 weeks) of either active high-frequency rTMS or sham stimulation. Participants will regularly complete measures to evaluate changes in pain severity and interference. The primary clinical outcome measures will be pain severity and interference scores on the Brief Pain Inventory (BPI). Additionally, participants will undergo MRI/MRS scans before and after the 5 weeks of rTMS to evaluate target engagement and help elucidate the potential mechanism of action of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic pain (back pain, osteoarthritis, complex regional pain syndrome, phantom limb pain, thalamic pain, pain related to injury of nerve plexus/plexi, or neuropathic facial pain).
2. Able to give informed consent, and comply with study procedures.
3. Opioid use disorder, moderate or severe.
4. Enrolled in methadone maintenance treatment program for at least 2 months and at least 1 month on a stable dose of methadone (up to 300mg/day).

Exclusion Criteria:

1. Medical conditions that preclude rTMS, including glaucoma, increased intracranial pressure, cardiac disease, migraine disorder, cerebral vascular events (CVA, TIA) any brain lesions (such multiple sclerosis),or seizure disorders.
2. Meet DSM-5 criteria for major psychiatric illness, such as bipolar disorder, major depression (severe), suicidal thoughts, mania, or psychosis, that would interfere with participation or pose a risk for rTMS.
3. Cognitive disorder.
4. Currently pregnant.
5. Metal implants or paramagnetic objects contained within the body which may interfere with the MRI scan, as determined in consultation with a neuroradiologist and according to the guidelines set forth in the following reference book commonly used by neuroradiologists: "Guide to MR procedures and metallic objects" Shellock, PhD, Lippincott-Raven press, NY 1998.14. This includes metal or shrapnel or bullet in the head or body, including metal shavings.
6. Subjects with positive responses to the Transcranial Magnetic stimulation Adult safety screen (TASS).
7. Currently taking a medication known to increase the risk of seizure.
8. Subjects with claustrophobia making them unable to tolerate MRI scanning.
9. Subjects involved in litigation regarding injury or worker's compensation benefits.
10. Subjects with a diagnosis of vasculitis, peripheral vascular disease, peripheral neuropathy, small-fiber neuropathy, or fibromyalgia.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Martinez, MD, Principal Investigator — New York Sate Psychiatric Institute / Columbia University; Derek Blevins, MD, Principal Investigator — New York State Psychiatric Institute / Columbia University
Locations (1):
- Substance Treatment and Research Service (STARS), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active rTMS Stimulation | Sham rTMS Stimulation
Started | 4 | 3
Completed | 1 | 3
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS Stimulation | Sham rTMS Stimulation | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (6) | 39 (5) | 37 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 2 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Ability to Recruit and to Have Participants Complete the Study
Description: Number of participants with chronic pain and comorbid psychiatric disorders who complete 60% of sessions.
Time Frame: 3 months
Population: In this feasibility study all participants were included in determining feasibility.
Measure: Count of Participants; unit: Participants
Arm/Group | Active rTMS Stimulation | Sham rTMS Stimulation
Number analyzed (Participants) | 4 | 3
Participants | 4 | 3

ADVERSE EVENTS:
Time Frame: Participants were followed for 9 weeks.
Arm/Group | Active rTMS Stimulation | Sham rTMS Stimulation
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 2/4 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active rTMS Stimulation (N=4) | Sham rTMS Stimulation (N=3)
headache (Nervous system disorders) | 2 (2) | 2 (2) — Mild headache reported with TMS (both groups)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT02687360/Prot_SAP_000.pdf